CLINICAL TRIAL: NCT06626802
Title: Intralesional Steroid Injection Versus Topical Mitomycin-C Use in Pediatric Benign Recurrent Esophageal Stricture: A Randomized Control Trial
Brief Title: Steroid Versus Mitomycin-C Use in Pediatric Benign Recurrent Esophageal Stricture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Collaborators: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Tehreem Fatima, Senior Registrar, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PedEsoStricture
Record Dates: First submitted 2024-09-24; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Stricture
Keywords: Esophageal stricture; Mitomycin; Triamcinolone; Dysphagia
MeSH Terms: conditions — Esophageal Stenosis; Deglutition Disorders | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Mitomycin (Experimental): Patients in Group A will be treated with esophageal dilation with a CRE balloon. After adequate dilation of stricture, injection Mitomycin will be applied to the narrowest portion of the stricture. It will be applied in a dose of 1ml (0.4mg/ml); after dividing in to four aliquots, each aliquot will be applied to to one of the four quadrants.
  Interventions: Procedure: Balloon Dilation + Topical Mitomycin
- Group B: Triamcinolone (Experimental): Patients in Group B will be treated with esophageal dilation with a CRE balloon. After adequate dilation of stricture, Triamcinolone injection will be injected into the narrowest portion of the stricture, using a sclerotherapy injector. Injection triamcinolone will be used in a dose of 1ml (40mg/ml). It will be divided in to four aliquots; each aliquot will be injected in to each of the four quadrants.
  Interventions: Procedure: Balloon Dilation + Injection Triamcinolone

INTERVENTIONS:
Procedure: Balloon Dilation + Topical Mitomycin — Patients with recurrent esophageal strictures in Group A will undergo endoscopy and balloon dilation with a CRE balloon, followed by injection Mitomycin applied topically at stricture site (post dilation)
  Arms: Group A: Mitomycin
Procedure: Balloon Dilation + Injection Triamcinolone — Patients with recurrent esophageal strictures in Group B will undergo endoscopy and balloon dilation with a CRE balloon, followed by injection Triamcinolone, injected with a sclerotherapy injector, at stricture site (post dilation)
  Arms: Group B: Triamcinolone

SUMMARY:
To compare the efficacy of steroid injection versus topical mitomycin-C in the treatment of pediatric benign recurrent esophageal strictures. The rationale for this study is to compare the two therapeutic options in order to measure their effectiveness, in terms of improvement of Dysphagia Severity Score (DSS).

DETAILED DESCRIPTION:
After taking approval from the Institutional Review Board of the university; and taking the informed consent from parents, patients fulfilling the inclusion and exclusion criteria will be enrolled in the study. They will be then randomly allocated into two groups; group A and group B. Patients in Group A will be treated with esophageal dilation with a CRE balloon (controlled radial expansion balloon). After adequate dilation of stricture, injection Mitomycin will be applied to the narrowest portion of the stricture. Patients in Group B will be treated with esophageal dilation with a CRE balloon in the same manner. After adequate dilation of stricture, Triamcinolone injection will be injected into the narrowest portion of the stricture, using a sclerotherapy injector. Dysphagia Severity Score will be noted at start of intervention, at 2 weeks after intervention and at 6 weeks post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients up to 16 years of age belonging to both genders
* Patients with single esophageal stricture
* Patients with benign recurrent esophageal strictures
* Patients with any etiology for esophageal stricture including; post-corrosive, congenital, post-anastomotic and eosinophilic.

Exclusion Criteria:

* Patients unfit for anesthesia and/or hemodynamic instability
* Patients with hemostatic disorder (platelets <50,000 or international normalized ratio >1.5)
* Patients who have undergone esophageal surgery in last one month
* Patients with complications such as; stricture perforation, signs of air leak or mediastinitis
* Those with hypersensitivity to Mitomycin- C
* Patients with multiple strictures

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness measured in terms of improvement in Dysphagia Severity Score (DSS) | 6 weeks
  Patients in both groups (group A and group B) will be followed and mean dysphagia severity score will be noted at 0, 2 and 6 weeks of intervention in both the groups. Improvement in dysphagia will be monitored via a validated Dysphagia Severity Score (DSS). It is as follows:
  0 Able to eat normal diet/no dysphagia
  1. Able to swallow some solid foods
  2. Able to swallow only semi solid foods
  3. Able to swallow liquids only
  4. Unable to swallow anything/total dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Fatima, FCPS, MRCPCH, Principal Investigator — University of Child Health Sciences, Lahore
Locations (1):
- Children Hospital and University of Child Health Sciences Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarma MS, Tripathi PR, Arora S. Corrosive upper gastrointestinal strictures in children: Difficulties and dilemmas. World J Clin Pediatr. 2021 Nov 9;10(6):124-136. doi: 10.5409/wjcp.v10.i6.124. eCollection 2021 Nov 9. PMID 34868889
- [Background] Al Sarkhy AA, Saeed A, Hamid YH, Al Asmi MM, Altokhais TI, Ullah AA, Assiri AM. Efficacy and safety of endoscopic dilatation in the management of esophageal strictures in children. Saudi Med J. 2018 Aug;39(8):787-791. doi: 10.15537/smj.2018.8.22845. PMID 30106416
- [Background] Boregowda U, Goyal H, Mann R, Gajendran M, Patel S, Echavarria J, Sayana H, Saligram S. Endoscopic management of benign recalcitrant esophageal strictures. Ann Gastroenterol. 2021;34(3):287-299. doi: 10.20524/aog.2021.0585. Epub 2021 Jan 27. PMID 33948052
- [Background] Ravich WJ. Endoscopic Management of Benign Esophageal Strictures. Curr Gastroenterol Rep. 2017 Aug 24;19(10):50. doi: 10.1007/s11894-017-0591-8. PMID 28840483
- [Background] Shahein AR, Krasaelap A, Ng K, Bitton S, Khan M, Manfredi MA, Lerner DG. Esophageal Dilation in Children: A State of the Art Review. J Pediatr Gastroenterol Nutr. 2023 Jan 1;76(1):1-8. doi: 10.1097/MPG.0000000000003614. Epub 2022 Sep 19. PMID 36122370
- [Background] Divarci E, Celtik U, Dokumcu Z, Ozcan C, Erdener A. The Efficacy of Intralesional Steroid Injection in the Treatment of Corrosive Esophageal Strictures in Children. Surg Laparosc Endosc Percutan Tech. 2016 Dec;26(6):e122-e125. doi: 10.1097/SLE.0000000000000351. PMID 27846162
- [Background] Dasari CS, Jegadeesan R, Patel HK, Desai M, Aziz M, Thoguluvachandrasekar V, Duvvuri A, Kohli DR, Repici A, Siersema PD, Sharma P. Intralesional steroids and endoscopic dilation for anastomotic strictures after esophagectomy: systematic review and meta-analysis. Endoscopy. 2020 Sep;52(9):721-726. doi: 10.1055/a-1172-5975. Epub 2020 May 25. PMID 32450581
- [Background] Mendez-Nieto CM, Zarate-Mondragon F, Ramirez-Mayans J, Flores-Flores M. Topical mitomycin C versus intralesional triamcinolone in the management of esophageal stricture due to caustic ingestion. Rev Gastroenterol Mex. 2015 Oct-Dec;80(4):248-54. doi: 10.1016/j.rgmx.2015.07.006. Epub 2015 Oct 9. English, Spanish. PMID 26455483